CLINICAL TRIAL: NCT00450307
Title: 3F8 Antibody Dose Escalation Plus Granulocyte-Macrophage Colony-Stimulating Factor in High-Risk Neuroblastoma: A Phase I Trial
Brief Title: Monoclonal Antibody 3F8 and GM-CSF in Treating Young Patients With High-Risk, Refractory or Relapsed Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-015; MSKCC-05015
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma; stage 4S neuroblastoma; disseminated neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — humanized 3F8 anti-GD2 monoclonal antibody; sargramostim

ARMS (1):
- 3F8 and GM-CSF (Experimental): One cycle has 5 days of 3F8 treatment. Each day, patients receive GM-CSF subcutaneously ~1.5 hr before the start 3F8 infusion. To limit side-effects, patients receive analgesics, antihistamines, and a small dose (IV, over ~5 minutes) of heat-modified 3F8. Cycles can be repeated after a 2-4 week interval, up to a total of two cycles.
  Interventions: Biological: monoclonal antibody 3F8; Biological: sargramostim

INTERVENTIONS:
Biological: monoclonal antibody 3F8
Biological: sargramostim

SUMMARY:
RATIONALE: Monoclonal antibodies, such as 3F8, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving monoclonal antibody therapy together with GM-CSF may be an effective treatment for neuroblastoma.

PURPOSE: This phase I trial is studying the side effects and best dose of monoclonal antibody 3F8 when given together with GM-CSF in treating young patients with high-risk, refractory or relapsed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of monoclonal antibody 3F8 when administered with sargramostim (GM-CSF) in young patients with high-risk, refractory or relapsed neuroblastoma.
* Assess anti-neuroblastoma effects of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of monoclonal antibody 3F8.

Patients receive sargramostim (GM-CSF) subcutaneously once daily on days -5 to 11 and monoclonal antibody 3F8 IV over 30 minutes on days 0-4 and 7-11. Treatment repeats every 4-6 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of monoclonal antibody 3F8 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of NB as defined by international criteria,45 i.e., histopathology (confirmed by the MSKCC Department of Pathology) or BM metastases plus high urine catecholamine levels.
* Patients must have refractory or relapsed high-risk NB (including MYCNamplified stage 3/4/4S and MYCN-nonamplified stage 4 >18 months old) resistant to standard therapy.
* Prior treatment with 3F8 is allowed.
* Age <21 years.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Existing major organ dysfunction should be grade 2 or less, with the exception of myelosuppression (neutrophil count >500/ul and platelet count >10,000/ul are acceptable), alopecia, hearing loss. Patient cannot be taking antihypertensive medication.
* History of allergy to mouse proteins.
* Active life-threatening infection.
* Human anti-mouse antibody (HAMA) titer >1000 ELISA units/ml.
* Prior treatment with 3F8 is NOT an exclusion criterion.
* Inability to comply with protocol requirements.
* Pregnant women are excluded for fear of danger to the fetus. Therefore negative pregnancy test is required for all women of child-bearing age, and appropriate contraception is used during the study period.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2005-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of monoclonal antibody 3F8 | 2 years
Anti-neuroblastoma effects of monoclonal antibody 3F8 and sargramostim (GM-CSF) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian H. Kushner, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Kushner BH, Kramer K, Modak S, Cheung NK. Successful multifold dose escalation of anti-GD2 monoclonal antibody 3F8 in patients with neuroblastoma: a phase I study. J Clin Oncol. 2011 Mar 20;29(9):1168-74. doi: 10.1200/JCO.2010.28.3317. Epub 2011 Feb 22. PMID 21343563